CLINICAL TRIAL: NCT01882179
Title: MINeralocorticoid Receptor Antagonist Pretreatment to MINIMISE Reperfusion Injury After ST-Elevation Myocardial Infarction (STEMI)
Brief Title: Early Mineralocorticoid Receptor Antagonist Treatment to Reduce Myocardial Infarct Size
Acronym: MINIMISE-STEMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12/0533
Record Dates: First submitted 2013-06-17; First posted 2013-06-20 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-05

CONDITIONS: ST-elevation Myocardial Infarction
Keywords: Reperfusion injury; myocardial infarct size; MRI; spironolactone
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Intravenous saline bolus prior to PPCI followed by oral placebo for 3 months
  Interventions: Drug: placebo
- Mineralocorticoid receptor antagonist (Active Comparator): 1st dose (day 0) given i.v. (potassium-canrenoate), before primary PCI day 1 - 12 weeks: spironolactone 25mg daily, which is uptitrated to 50mg daily after 2 weeks, if possible
  In case the LVEF <40% on baseline MRI and the patient shows signs of heart failure or is diabetic, the patient will receive open label eplerenone instead of the study drug, according to current guidelines.
  Interventions: Drug: Mineralocorticoid receptor antagonist potassium-canrenoate

INTERVENTIONS:
Drug: Mineralocorticoid receptor antagonist potassium-canrenoate
  Arms: Mineralocorticoid receptor antagonist
Drug: placebo
  Arms: Placebo

SUMMARY:
Heart attacks, or myocardial infarcts, are a major cause of death and disability in the UK. Immediate unblocking of the obstructed heart vessel with a balloon catheter and implantation of a mesh scaffold (stent) in heart centers is warranted in these patients. Morbidity and mortality in this patient group is related to the infarct size. Therefore, there is a need to discover novel therapeutic agents which reduce myocardial infarct size and preserve the contractile heart function.

Large trials involving several thousand patients have demonstrated a survival benefit in patients with impaired heart function due to a heart attack, who received a mineralo-corticoid receptor antagonist (MRA, drug name: spironolactone). In these trials patients received the drug late, 3-14 days after the heart attack.

Our proposal is to investigate whether MRA therapy administered intravenously prior to unblocking an occluded heart vessel, can reduce infarct size and as such can prevent long term sequelae of heart attacks.

150 patients admitted to 4 tertiary care hospitals (Heart Hospital London, London Chest, Essex Cardiothoracic Center and Leeds General Infirmary) for heart attack will be randomly assigned to receive MRA treatment or placebo. The first dose of the MRA will be applied intravenously immediately in the catheter suite, even before re-opening of the occluded vessel. From the second day on, patients will be prescribed oral MRA treatment, as a pill, for a total of three months. Before hospital discharge and after three months, a magnetic resonance image (MRI) of the heart will accurately investigate the evolution of infarct (scar) size and the contractile heart function and compare the group of patients who received the MRA drug versus the placebo control group. Of note, patients with an ejection fraction <40% AND signs of heart failure OR diabetes will go on open label eplerenone according to current guidelines, instead of the study drug.

This study will give first evidence, if very early MRA treatment improves heart function and should be used as early as possible for treatment of patients after a heart attack.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for entry into trial

* Patients >18 years
* Patients presenting with acute STEMI (as assessed by 12 lead ECG; ST segment elevation ≥2 mm (0.2 mV) in 2 or more contiguous precordial leads or ≥1mm (0.1mm) in 2 or more adjacent limb leads).
* Presentation within 12 hours after symptom onset

Inclusion criteria for randomization (assessed in catheter laboratory)

* Angiographically proven proximal occlusion (TIMI 0) of a major coronary vessel (LAD, LCX, RCA).
* Normal potassium (<5.0 mmol/l)

Exclusion Criteria:

* Patients with known LVEF ≤40%
* Participation in another trial
* Cardiogenic shock (positive shock index OR need for catecholamine support OR systolic blood pressure < 90 mmHg)
* Killip class > 2
* Prior myocardial infarction
* Known compromised renal function (eGFR < 30 ml/min/1.73 m2) or potassium > 5.0 mmol/l
* Current treatment with mineralocorticoid receptor antagonists
* Pregnant or lactating females
* Allergies to IMP or its excipients
* Known contraindication to cardiac magnetic resonance imaging (MRI) such as significant claustrophobia, severe allergy to gadolinium chelate contrast, , presence of MRI contraindicated implanted devices (eg, pacemaker, implanted cardiac defibrillator, cardiac resynchronization therapy device, cochlear implant), imbedded metal objects (eg, shrapnel), or any other contraindication for cardiac MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Myocardial infarct (MI) size, as assessed by cardiac magnetic resonance imaging | 12 weeks after STEMI

SECONDARY OUTCOMES:
Markers of myocardial reperfusion injury | 48 hours
  TIMI flow post-PPCI, ST-segment resolution post-PPCI
Microvascular obstruction on cardiac MRI | 1-3 days after STEMI
  hypodense area of late gadolinium enhancement
Myocardial salvage | 12 weeks
  Area at risk assessed by T2 weighted imaging subtract final MI size
Acute myocardial infarct size | 1-3 days
  serum biomarkers: hsTnT, CK-MB, CK and cardiac MRI: late gadolinium enhancement
LV remodelling | 12 week cardiac MRI scan
  LV end-diastolic and end-systolic volumes, LV ejection fraction, LV mass and wall-thickness
Clinical outcome measures | 12 weeks
  cardiovascular death, non-fatal myocardial infarction, revascularisation, hospitalisation for heart failure, hyperkalemia, deterioration of kidney function, need for dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Derek J Hausenloy, PhD, Study Director — University College London, Hatter Cardiovascular Institute; Georg M Fröhlich, MD, Study Chair — University College London, The Heart Hospital; Pascal Meier, MD, Principal Investigator — University College London, The Heart Hospital; Reto Gamma, MD, Principal Investigator — Basildon and Thurrock University Hospitals; Anthony Mathur, PhD, Principal Investigator — London Chest Hospital; John Greenwood, MD, Principal Investigator — Leeds General Infirmary
Locations (4):
- United Kingdom (4):
  - Cardiothoracic Center - Basildon and Thurrock University Hospitals, Basildon, Essex
  - London Chest Hospital, London, London
  - Heart Hospital London, London, London
  - Leeds Genereal Infirmary, Leeds

REFERENCES:
- [Background] Pitt B, Remme W, Zannad F, Neaton J, Martinez F, Roniker B, Bittman R, Hurley S, Kleiman J, Gatlin M; Eplerenone Post-Acute Myocardial Infarction Heart Failure Efficacy and Survival Study Investigators. Eplerenone, a selective aldosterone blocker, in patients with left ventricular dysfunction after myocardial infarction. N Engl J Med. 2003 Apr 3;348(14):1309-21. doi: 10.1056/NEJMoa030207. Epub 2003 Mar 31. PMID 12668699
- [Background] Zannad F, McMurray JJ, Krum H, van Veldhuisen DJ, Swedberg K, Shi H, Vincent J, Pocock SJ, Pitt B; EMPHASIS-HF Study Group. Eplerenone in patients with systolic heart failure and mild symptoms. N Engl J Med. 2011 Jan 6;364(1):11-21. doi: 10.1056/NEJMoa1009492. Epub 2010 Nov 14. PMID 21073363
- [Background] Pitt B, Zannad F, Remme WJ, Cody R, Castaigne A, Perez A, Palensky J, Wittes J. The effect of spironolactone on morbidity and mortality in patients with severe heart failure. Randomized Aldactone Evaluation Study Investigators. N Engl J Med. 1999 Sep 2;341(10):709-17. doi: 10.1056/NEJM199909023411001. PMID 10471456
- [Background] Schmidt K, Tissier R, Ghaleh B, Drogies T, Felix SB, Krieg T. Cardioprotective effects of mineralocorticoid receptor antagonists at reperfusion. Eur Heart J. 2010 Jul;31(13):1655-62. doi: 10.1093/eurheartj/ehp555. Epub 2009 Dec 21. PMID 20028693